CLINICAL TRIAL: NCT03243110
Title: The Economic Burden of Asthma in Canada
Acronym: PopData
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Mark Fitzgerald, Professor, University of British Columbia
Other Study IDs: H10-01542
Record Dates: First submitted 2017-08-03; First posted 2017-08-08 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Breath Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Asthmatics requiring breathing test: Participants must have had a diagnosis of asthma by a physician. The participant must have had a self-reported health care interaction related to asthma (physician visit, ED visit, hospitalization) in the past 5 years.
  Participants must be 1 to 85 years old.
  Interventions: Diagnostic Test: breathing test

INTERVENTIONS:
Diagnostic Test: breathing test — Spirometry is a non-invasive means of measuring lung function: The participant is asked to take a deep breath and then exhale into the sensor as hard and as long as possible. Soft nose clips may be used to prevent air escaping through the nose. If the participant does not show a definitive diagnosis of asthma, a methacholine challenge test will be performed to elicit bronchoconstriction in participants. In methacholine challenge test, the participant breaths in standardized dose of nebulized methacholine again. Methacholine challenge test is widely accepted and standardized method for assisting the diagnosis of asthma and there will be no experimental altercation in the method methacholine challenge is performed.

SUMMARY:
The study will consist of three phases: Phase A: General population survey for estimation of the prevalence of asthma, and prospective collection of resource utilization and quality-of-life data for 12 months, Phase B: comparison of healthcare resource usage collected prospectively to the data collected using administrative data in the population recruited in Phase A, and Phase C: Economic modeling of asthma to extrapolate the findings across Canada and into the future years.

DETAILED DESCRIPTION:
Phase A: This phase will be a prospective cohort study of randomly chosen residents of two census subdivisions of BC with a self-reported physician diagnosis of asthma. The study participants will be recruited via landline and cell phone-based random digit dialing across two regions in British Columbia: the Census Sub-Division of the city of Vancouver and the Census Division of Central Okanagan. The target area was chosen based on Census Sub-Division as it provides a clear definition of the target population for whom demographic and socioeconomic data is available through national and provincial census and surveys. The Okanagan Census Sub-Division was particularly chosen as it provides data on both urban and rural populations (18.6% rural population in 2006). According to 2006 census profile, the population of these two Census Sub-Divisions is, respectively, 578,041 and 162,276. Accordingly, about 78% of participants would be recruited from Vancouver, and 22% from Okanagan. The study will randomly sample participants from all the area codes in these regions. The target population will include household residents residing in telephone exchanges within the target Census Sub-Divisions. Random digit dialing will be geographically stratified with an associated sample weight that will approximate a probability sample of the individuals in the population. Previous studies have shown that acceptably high response rates can be achieved among Canadian participants with asthma.

Random digit dialing samples have been shown to be more representative than population samples drawn using alternative methods such as telephone directories or electronic white pages. However, random digit dialing is not free of bias. Non-random non-response is an issue, and it has been shown that reducing the non-response rate may directly reduce non-response bias. Non-responders in random digit dialing may not have been contacted because the non-responders work multiple minimum-wage jobs. The investigators will place multiple calls and leave messages on answering machines. Random digit dialing is also subject to no-telephone bias - households without telephones are out of reach by random digit dialing, and the households without telephones probably differ in socioeconomic status than the overall population. However, for the urban, suburban, and semi-rural sub-populations within British Columbia, telephone coverage is almost universal.

Inclusion of cell phones in random digit dialing is an attempt to mitigate such biases and increase the fraction of population covered by sampling. More importantly, the inclusion of cell phones is likely to result in inclusion of participants that might be absent from landline random digit dialing (younger and more educated groups) thus mitigating the sampling bias of random digit dialing. Cell phone random digit dialing is an active area of research and it is too soon to know with confidence what should and should not be regarded as a "Best Practice". For inclusion of cell phones in random digit dialing, the investigators will use the "Screening Approach". In this approach the interview is only conducted with participants sampled via the cell phone frame who do not have a landline, thus excluding numbers from the cell phone sample in the overlap (i.e., screening out the participants with both a cell phone and a landline). In this alternative sampling design, participants who have at least one household landline telephone and use at least one cell phone would be eligible for inclusion only from the landline frame. This decreases the bias due to higher probability of sampling from households who have both a landline and cell phone.

The study will employ the Waksberg method of random digit sampling. In this method, all telephone numbers are initially split into blocks of equal size, called "primary sampling units". The primary sampling unit will be a mixture of landlines and cell phones. One randomly selected telephone number is called from each selected primary sampling unit. When a residential connection is reached in the first stage, the primary sampling unit qualifies for inclusion in the second stage.

Respondents will be asked the following question: "Is there a member of the household between ages of 1 to 85 who has had asthma ever diagnosed by a physician". If the response is affirmative the study assistant will ask if the participant in question can continue the conversation directly (parents in case of children). Eligible participants (or in the case of children their parents or guardians) will be informed of the objectives of the study, verbally consented, and then screened for eligibility based on age and history of asthma. Participants who meet eligibility criteria and verbally consent over the phone will be asked to come to the study laboratory (one at Vancouver and one at Kelowna, corresponding to the two Census Sub-Divisions) and the participant will receive a detailed explanation of the study and the study consent form at that time.

All participants who provide signed consent will then proceed to spirometry (simple spirometry without bronchodilator response) and study data collection. After the baseline visit, participants enter a 12-months period of follow-up with visits at months 3, 6, 9, and 12. Participants will be asked to attend one of the study centres and data on the quality of life and asthma-related resource utilization will be gathered. On the final visit, participants will undergo spirometry for objective diagnosis of asthma with possible methacholine challenge test for the participants whose asthma cannot reliability be included or excluded.

Phase B: In this phase of the study, health records of participants who have participated in the phase A of the study for the entire follow-up period and the 12 months period prior to the participants' enrolment will be retrieved from the BC Linked Health Database. In addition, the investigators will identify cases of asthma in the entire British Columbia population based on the administrative data for the same period of time. The BC Linked Health Database is a longitudinal administrative health care database containing participant-specific, anonymized health data from 1985 onwards on British Columbia's 4 million residents with health insurance. Records will be matched based on participants' unique Personal Health number and hence the matching will be almost completely accurate. Data extracted from the BC Linked Health Database will include Medical Services Plan data, which encompass fee-for-service physicians, the Discharge Abstracts Database of hospital inpatient separation records, as well as records of death certificates. Prescription drug use will be determined from the BC Pharmanet database. This is a population-based prescription drug database that captures essentially all dispensing episodes by outpatients residing in the province on a prescription-by-prescription basis (regardless of funding source)..

One request thought the British Columbia ministry of health (personal communication with Data Stewardship Secretariat) is required to retrieve data on the study participants as well as cases of asthma across the entire province, without additional cost for the latter group. The investigators will use this opportunity to retrieve data on cases of asthma in the entire province and compare different aspects of resource utilization between objectively verified cases of asthma and the data retrieved using a case definition algorithm on an administrative database. Such data will be used to retrospectively estimate the direct costs of asthma during the follow-up and in the 12 months prior to the enrolment in the study. The direct medical costs calculated in this way will be compared with the direct costs calculated in the prospective phase of the study. In addition, the investigators will examine the representativeness of the sample population by comparing the participant's health records with case of asthma in British Columbia identified through the BC Linked Health Database. Given the objective validation of the diagnosis of asthma at the end of the follow-up period in Phase A, the investigators will also be able to explore the sensitivity of existing case ascertainment algorithms based on administrative data at levels of severity and control.

Phase C: Economic model of asthma: The data collected from participants during this study will be extrapolated to the population of British Columbia and Canada by appropriate adjustment for demographic and socioeconomic differences and reported prevalence of asthma in the country. The data will also be used to populate a Markov model of asthma to project the burden of asthma for the next 10 years. The Markov model of asthma will extend the model previously developed by Price et al. However, the investigators will model all 4 states of severity as defined by the Global Initiative in Asthma and whether at each year the participant's symptoms are controlled or uncontrolled. The Markov model will hence consist of 8 states (plus state of death) for all permutations of levels of severity and control. The model will also incorporate both the steady-state of chronic asthma and the acute state associated with an asthma exacerbation. Whenever possible, the investigators will estimate the parameters of the model from the cohort of participants in the Phase A and B of the study. This will include the initial distribution of individuals according to levels of severity and control, and the quality of life weights and annual direct and indirect costs estimated from the statistical analysis of the cohort data. The long term transition probabilities among levels of severity and control cannot reliably be estimated given the short follow-up of the participants in this study. The investigators will use values estimated from the literature for these and other components of the model.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must state that they have had a diagnosis of asthma by a physician. In addition, the patient must have had a self-reported health care interaction related to asthma (physician visit, ED visit, hospitalization) in the past 5 years.
2. Patient must be 1 to 85 years old.

   -

Exclusion Criteria:

1. Patients unable to provide informed consent due to language difficulties or cognitive impairment.
2. Patients who have a greater than 10 pack-year smoking history (this will exclude patients with possible COPD).
3. Patients who know that they will be moving out of the province within 12 months of study entry.
4. Patients in whom metacholine challenge test is contraindicated due to non-asthma-related reasons (e.g. patients with cerebral aneurysm, pregnant and breastfeeding participants).

   -

Ages: 1 Year to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Phase A of the study will be based on the survey of the general population (1-85 y/o) of two well-defined target areas and recruitment of those with a self-reported physician diagnosis of asthma. Phase B of the study is the retrospective elicitation of the health record of participants. In Phase C of the study builds upon the data of Phase A and B and other published studies to extrapolate the results to the Canadian population for the next 10 years, as such it does not involve direct population sampling.
Sampling Method: Non-Probability Sample
Enrollment: 613 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Costs of asthma in BC and Canada per patient | September 2013
  Costs per patients will be calculated by multiplying the amount of healthcare resources used by the corresponding unit costs. The investigators will adjust all unit costs to 2010 Canadian dollar according to the medical care component of the Consumer Price Index(42). The lowest price for available (generic drugs if exists) versions of medications will be used based on province-specific data.

SECONDARY OUTCOMES:
Calculating quality of life of participants with asthma using the Asthma Quality of Life Questionnaire | January 2017
  The investigator will report mean from the Asthma Quality of Life Questionnaire (Pediatric Asthma Quality of Life Questionnaire in children) for each participant. The mean Asthma Quality of Life Questionnaire score for baseline and each follow-up visit among all participants will also be calculated. The investigator will use a linear mixed model (with a random effect parameter for each participant) to calculate the rate of change in Asthma Quality of Life Questionnaire over the study period.
Calculating quality of life of participants with asthma using the EuroQol's EQ-5D Questionnaire | February 2017
  The investigator will report mean from the EuroQol's EQ-5D data. Based on the available EuroQol's EQ-5D responses for each participant, the investigator will calculate the Quality Adjusted Life Years for each participant, assuming linear change in EuroQol's EQ-5D scores between successive measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Mohsen Sadatsafavi, MD,Ph.D, Study Chair — University of British Columbia

IPD SHARING:
Plan to Share IPD: Undecided